CLINICAL TRIAL: NCT06720818
Title: Mucosal Associated Invariant T Cell During Viral Pneumonia and Acute Respiratory Distress Syndrome
Acronym: MAIT-VECTORS
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: DR230303 - MAIT-VECTORS
Record Dates: First submitted 2024-11-25; First posted 2024-12-06 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Viral Pneumonia; Acute Respiratory Distress Syndrome (ARDS)
Keywords: Mucosal Associated Invariant T cell; physiopathology; immune response
MeSH Terms: conditions — Pneumonia, Viral; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and respiratory samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Viral pneumonia, including SARS-CoV-2 and influenza A virus (IAV), can culminate in acute respiratory distress syndrome (ARDS), a severe form of respiratory failure with high mortality. Uncontrolled local inflammatory response and impaired tissue repair are hallmarks of ARDS. However, lack of in-depth understanding of the immunopathology lead to limited identification of potential 'endotypes' who may benefit from individualized targeted therapies. Mucosal Associated Invariant T (MAIT) cells represent a peculiar lineage of T cells with a wide panel of effector functions. Thus, they emerge as potential key players and appealing targets in ARDS through their potent abilities to modulate immune response at barrier sites and promote tissue repair. Recent data from the investigators and others indicated that MAIT cells are highly activated in patients with Sars-Cov-2 and IAV ARDS, but the associated activation mechanisms and precise functions remain unknown.

In this context, the investigators aim at investigating the implication and potential harnessing of MAIT cells in severe viral pneumonias and associated ARDS by with a dedicated clinical study. First, the investigators will perform a comprehensive and longitudinal phenotyping of immune response during viral pneumonia-induced ARDS, including MAIT cells, in blood -and airway compartment for mechanically ventilated patients. To provide more insight into specificity of virally induced pneumonia and ARDS, longitudinal phenotyping of immune response of patients with bacterial pneumonia, and control patients with unrelated ARDS (severe trauma, pancreatitis or major surgery) will also be performed.

DETAILED DESCRIPTION:
Viral pneumonias, notably those caused by Sars-CoV-2 and influenza, are important threats for humans. Both viral infection and subsequent activation of the immune system result in lung injury. In severe cases, disruption of the lung alveolo-capillary membrane and associated edema impair gas exchanges, requiring admission in intensive care unit (ICU) and respiratory support. Uncontrolled local immune response, non-resolving inflammation and impaired tissue repair may develop in few days and perpetuate respiratory failure, forming the so-called 'Acute Respiratory Distress Syndrome' (ARDS), which culminates with a mortality rate close to 40%. Pathophysiology of ARDS remains poorly understood, which may explain the absence of immunomodulatory treatments despite numerous clinical trials, except for steroids in severe COVID-19. To develop new treatments, the investigators need to dissect the immunopathology of ARDS with new approaches and provide pathophysiological 'endotypes' to lead to future precision-medicine clinical trials1. Here, the investigators will investigate implication and therapeutic use of Mucosal Associated Invariant T (MAIT) cells. MAIT cells recently emerged as key-players in immune responses at barrier sites, including the lungs, where they modulate local immune responses and promote tissue repair. Given their rapid and wide effector potential, MAIT cells are particularly relevant in acute conditions such as ARDS. Interestingly, MAIT cells protect against lethal influenza infection in mouse models. In patients, MAIT cells are activated and their frequency is decreased in blood during severe bacterial and viral infections. In severe COVID-19 patients, the investigators and others showed that MAIT cells from blood and airways were strongly activated. Our preliminary results in other infectious ARDS show high frequency of activated blood MAIT cells, but not in ICU patients admitted for other reason than pneumonia, suggesting that activation does not result from the acute critical condition. While the investigators observed that high activation of MAIT cells in blood was associated with positive clinical outcome, other studies observed a negative association. These discrepancies, probably linked to differences in severity between cohorts, also suggest that MAIT cell play versatile (potentially opposite) functions according to the context in severe viral pneumonias and associated ARDS.

Thus, determining how and when these potentially contrasted functions are set and controlled during ARDS is paramount to target MAIT cells for treatment. Hence, the investigators need to i) better characterize MAIT cell phenotype and functions throughout virally-induced ARDS in patients; ii) develop a mechanistic approach to explore MAIT cell functions and therapeutic manipulation in such settings.

The study will enroll 150 patients admitted in ICU for influenza and COVID-19 pneumonia, bacterial pneumonia, and control patients with unrelated ARDS (severe trauma, pancreatitis or major surgery). In parallel with comprehensive longitudinal clinical assessment, the investigators will assess MAIT cell frequency and activation marker expression (CD69, CD56, PD-1) in blood and airways. Analysis of the other immune lineages will generate a comprehensive map of the immune response in association with MAIT cell. Among each group, 'prototypical' patients will be selected based on their clinical outcome: rapidly recovering, prolonged ICU stay and death. Blood MAIT cell function and other main myeloid and lymphoid cells will be extensively characterized throughout the disease, by RNA sequencing and secretome analysis. Integrative analysis of these data will define the differentiation patterns of MAIT cells, their dynamic and considered location (blood versus airways). The analysis will also test the hypothesis for which patients with poor outcome and non-resolving ARDS have less tissue-repair oriented MAIT cells.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients admitted to critical care (Intensive Care Unit, Continuous Monitoring Unit, Intensive Care Unit) at the CHRU de Tours
* Patients admitted to critical care for one of the following reasons:

  * Acute community-acquired pulmonary infection (pneumonia),
  * Severe acute pancreatitis, with onset of ARDS criteria less than 48 hours ago,
  * Severe isolated head injury requiring invasive mechanical ventilation,
  * Severe burn defined by a burned surface area exceeding 20% and/or deep lesions exceeding 3% of the total body surface area, with the onset of ARDS criteria less than 48 hours ago,
  * Patient admitted to Intensive Care Medicine, requiring invasive mechanical ventilation,
  * Patient admitted to cardiac surgery for scheduled surgery for valve replacement and/or coronary artery bypass grafting, with inclusion the day before surgery,

Non-inclusion criteria :

* Patients with severe immunosuppression (impairing the ability to analyse the immune response, particularly T lymphocytes): active haematological malignancy, solid organ transplantation or bone marrow transplantation, systemic immunosuppressive treatment, ongoing chemotherapy (including immune checkpoint inhibitors).
* Person who has objected to data processing
* Patient under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to critical care units at the CHRU de Tours for different reasons
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
MAIT cells frequency during pneumonia and ARDS | Blood and airway (tracheal aspiration or bronchoalveolar lavage, for patients under mechanical ventilation) will be sampled and analyzed at inclusion, day 3, day 5 and every week until ICU discharge (with a maximum of 90 days in ICU after inclusion)
  MAIT cell frequency will be determined as % of CD3+ cells using flow cytometry techniques on biological samples obtained from samples done during routine care of patients included in the study (blood samples, and tracheal aspiration and broncho alveolar lavage for mechanically ventilated patients).

SECONDARY OUTCOMES:
Activation of MAIT cells during severe pneumonia and ARDS | Blood and airway (tracheal aspiration or bronchoalveolar lavage, for patients under mechanical ventilation) will be sampled and analyzed at inclusion, day 3, day 5 and every week until discharge (with a maximum of 90 days in ICU after inclusion).
  MAIT cell activation (expression of CD69, PD-1 and CD56), cytotoxicity markers (granzyme B, CD107a), and cytokine production (IL-17, IFNγ, IL-22) after PMA-ionmycin stimulation will be assessed using flow cytometry techniques on biological samples obtained from samples done during routine care of patients included in the study (blood samples, and tracheal aspiration and broncho alveolar lavage for mechanically ventilated patients) and ultimately expressed as % of activated MAIT cells.

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital, Tours, France

IPD SHARING:
Plan to Share IPD: Undecided